CLINICAL TRIAL: NCT05438927
Title: Early Supportive Care and Nutritional Support in Adults With Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Canopy Cancer Collective (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21795
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
Keywords: Nutritional Support
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Support (Experimental): Participants will receive individually tailored, bi-weekly nutrition counseling from a dietician via telehealth and remote monitoring through a smart phone app and wearable sensor to allow participants to log food intake while sharing data with a dietician
  Interventions: Behavioral: Fitbit Data Collection; Behavioral: Nutrition Counseling; Behavioral: Fact G Survey; Behavioral: General Anxiety Disorder (GAD)-7; Behavioral: Patient Health Questionnaire (PHQ)-9

INTERVENTIONS:
Behavioral: Fitbit Data Collection — Participants will log food intake while sharing their data with a dietician in real time for 12 weeks
Behavioral: Nutrition Counseling — Participants will receive individually tailored, biweekly nutrition counseling from a dietician via telehealth
Behavioral: Fact G Survey — Participants will take a survey at baseline and weeks 4,8,12 & 16. The questionnaire includes questions about participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher total score indicates better quality of life.
Behavioral: General Anxiety Disorder (GAD)-7 — Participants will take a survey at baseline and weeks 4,8,12 & 16. The questionnaire measures participants anxiety with a scale of 0=not at all, 3=Nearly everyday.
Behavioral: Patient Health Questionnaire (PHQ)-9 — Participants will take a survey at baseline and weeks 4,8,12 & 16. The questionnaire measures participants depression with a scale of 0=not at all, 3=Nearly everyday.

SUMMARY:
The purpose of the study is to assess the feasibility and patient satisfaction with the Support through Remote Observation and Nutrition Guidance (STRONG) program. The program provides nutrition and supportive care for participants living with pancreatic cancer who are receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Newly diagnosed metastatic or newly recurrent pancreatic cancer or locally advanced pancreatic cancer
* Planning to initiate chemotherapy under the guidance of Moffitt
* Able to speak and read English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g., psychosis, active substance abuse)
* Undergoing concurrent treatment for a second primary GI cancer
* ECOG status of 2 or greater
* Receipt of chemotherapy in the past 6 months for recurrent pancreatic cancer
* Use of parenteral or enteral nutrition
* Presence of malignant ascites
* The last two exclusion criteria were included because investigators do not anticipate that these patients would benefit from additional nutrition intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 50% of eligible participants are recruited
Data Collection - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 50% of participants submit study assessments
Participant Rating on Ease of Use for the Mobile Application - Usability | 12 Months
  The study will be deemed usable if ≥ 60% of participants rate the mobile application as easy-to-use for logging dietary intake

SECONDARY OUTCOMES:
Participant Compliance with Palliative Care Visits - Intervention Adherence | 12 Months
  Intervention adherence will be deemed successful if ≥ 60% of participants attend recommended palliative care visits (# of visits based on provider recommendation)
Participant Compliance with Dietician Visits - Intervention Adherence | 12 Months
  Intervention adherence will be deemed successful if ≥ 60% of participants meet with a dietician biweekly for 12 weeks
Participant Compliance with Dietary Log - Intervention Adherence | 12 Months
  Intervention adherence will be deemed successful if ≥ 60% of participants rack food intake for 8/12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi Tabriz, MD, PhD, Principal Investigator — Moffitt Cancer Center; Pamela Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE